CLINICAL TRIAL: NCT07104305
Title: Nudging and Relationship Building With Frequent Contact
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Deemed not feasible at current time.
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, David Ring, Professor, Dean associate of surgery department, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-07-0005
Record Dates: First submitted 2019-12-23; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Any Musculoskeletal Condition
Keywords: Musculoskeletal; Orthopedics; Mental health; Patient-Clinician relationship
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: New or return patients with some opportunity to better adapt to a long-standing or permanent symptoms will be randomized to a high-contact communication strategy agreed on by the clinician and patient or standard care (the patient initiates between visit contact as needed). The communication strategy may utilize text, email, portal, phone, video or other options as agreed on. The frequency will be at least once a week. All patients will complete a set of questionnaires at the end of the visit.
  At the end of the initial visit and 1 month after enrollment, people will be contacted by their method of choice to repeat the questionnaires.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care (No Intervention): Patients in this arm will receive the standard amount of contact with their clinician.
- High-contact communication strategy (Experimental): Patients will have contact with their clinician more frequently. The communication strategy may utilize text, email, portal, phone, video or other options as agreed on. The frequency will be at least once a week. All patients will complete a set of questionnaires at the end of the visit.
  Interventions: Behavioral: High-contact communication strategy

INTERVENTIONS:
Behavioral: High-contact communication strategy — Patients will have contact with their clinician more frequently. The communication strategy may utilize text, email, portal, phone, video or other options as agreed on. The frequency will be at least once a week. All patients will complete a set of questionnaires at the end of the visit.
  Arms: High-contact communication strategy

SUMMARY:
This study aims to test in what way a care strategy incorporating frequent contact can benefit patients with musculoskeletal condition that necessitates some adaptation and resiliency to symptoms and limitations that are expected to be either long-lasting or permanent.

Patients will be randomized into either group A, where they will receive the standard amount of contact with their clinician, or group B, in which they will have contact with their clinican more frequently.

The communication strategy may utilize text, email, portal, phone, video or other options as agreed on. The frequency will be at least once a week. All patients will complete a set of questionnaires at the end of the visit.

DETAILED DESCRIPTION:
Irregular and uncomfortable bodily symptoms are common. Most are well adapted in a healthy life. People seek care when a symptom becomes a concern. Even the effort to attend a routine healthy check-up is usually based on not wanting to miss anything, which is accompanied by at least a slight concern that a problem might be found. People that are seeking care are unsettled to some degree.

This unsettled feeling is often rooted in or worsened by unhelpful thoughts (less effective cognitive coping strategies). An example of a less effective cognitive coping strategy is rumination on worst-case thoughts (catastrophic thinking). The unsettled feeling is worse when thoughts are perceived as facts (cognitive fusion). Cognitive fusion is greater when people are under greater stress or distress.

Clinicians can help people feel better and do more by gently correcting these misconceptions. And when correction of misconceptions is to some degree at odds with a person's experience of reality, expert advice may seem impersonal, dismissive, and uncaring.

Adherence to medical expertise is enhanced by a trusting relationship with one's clinicians. There are several methods for nurturing a clinician-patient relationship. One is to make small agreements or compromises such as ordering a test that is not likely to yield useful information, has a small risk of harm, and uses resources and doing so in the context of efforts to move towards more effective cognitive coping strategies and greater self-efficacy. Another is to use educational tools such as decision aids to depersonalize the transfer of expertise. A third approach is use more frequent contact to deepen the relationship.

This study posits that establishing a frequent-contact plan with a patient that might benefit from a healthier inner narrative can improve health using few resources other than clinician time, with a good patient experience compared to the typical single or infrequent in person specialist office visits.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* New or return visit
* English or Spanish speaker
* A musculoskeletal condition that necessitates some adaptation and resiliency to symptoms and limitations that are expected to be either long-lasting or permanent

Exclusion Criteria:

* Cognitive dysfunction
* Language other than English or Spanish

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Guttman Satisfaction scale | 1 month after enrollment
  The Guttman Satisfaction Scale is a unidimensional questionnaire designed to measure the degree of patient satisfaction with the care they received. It consists of a series of hierarchically ordered yes/no items, with each successive item indicating a higher level of satisfaction. Total scores range from 0 to 7, with higher scores reflecting greater satisfaction, representing a better outcome.

SECONDARY OUTCOMES:
PROMIS Physical Function CAT | 1 month after enrollment
  Patient-perceived physical function will be assessed using the PROMIS® Computer Adaptive Test (CAT) Physical Function v2.0. This instrument dynamically selects items from a calibrated item bank to measure physical functioning, including mobility, self-care, and instrumental activities. Scores are reported as T-scores, standardized with a mean of 50 and a standard deviation of 10 in the general U.S. population. Higher scores indicate better physical function and therefore a better outcome.
Negative Pain Thoughts Questionnaire (NPTQ-4) | 1 month after enrollment
  A shortened version (4 items) of the Negative Pain Thoughts Questionnaire will be used to assess maladaptive cognitive coping strategies related to pain. Each item is rated on a 5-point Likert scale (0 = never to 4 = always), with total scores ranging from 0 to 16. Higher scores indicate more frequent negative pain-related thoughts, representing a worse outcome.
PROMIS Depression CAT | 1 month after enrollment
  Patient-perceived feelings of depression will be assessed using the PROMIS Depression Computer Adaptive Test (CAT) v1.2. This instrument selects items from a validated item bank to measure negative mood, loss of interest, and feelings of hopelessness. Scores are reported as T-scores, standardized with a mean of 50 and a standard deviation of 10 in the general U.S. population. Higher scores indicate greater depressive symptoms, representing a worse outcome.
Jefferson Scale of Patient's Perceptions of Physician Empathy (JSPPE) | 1 month after enrollment
  The Jefferson Scale of Patient's Perceptions of Physician Empathy includes five items rated on a 7-point Likert scale (1 = strongly disagree to 7 = strongly agree), with total scores ranging from 5 to 35. Higher scores indicate greater perceived physician empathy, representing a better outcome.
Communication effectiveness | 1 month after enrollment
  Two questions will be used to assess patient-perceived communication effectiveness, focusing on clarity, understanding, and responsiveness during the clinical interaction. Each item was rated on a 5-point Likert scale (1 = strongly disagree to 5 = strongly agree), with higher scores indicating more effective communication.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Health Austin (UTHA), Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No